CLINICAL TRIAL: NCT04215484
Title: Does Serum BNP Predict Abnormal Placental Invasion During Pregnancy
Brief Title: Placenta Accreta New Detection Procedure by Rapid Assessment of Serum BNP
Acronym: PANDORA
Status: Completed | Type: Observational
Sponsor: Ben marzouk Sofiene (Other)
Responsible Party: Sponsor-Investigator, Ben marzouk Sofiene, clinical associate professor, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Other Study IDs: BNP-ACCRETA
Record Dates: First submitted 2019-12-17; First posted 2020-01-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Placenta Accreta; Placenta Previa; Normal Pregnancy
Keywords: placenta previa; placenta accreta; BNP; cesarean section; pregnancy
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- P: P (previa) : pregnant women with placenta previa on ultrasound and no suggestive signs of placenta accreta
  Interventions: Diagnostic Test: serum BNP assessment
- I: I (abnormal placental Invasion) : pregnant women with placenta previa on ultrasound,and suggestive signs of placenta accreta on ultrasound with or without MRI
  Interventions: Diagnostic Test: serum BNP assessment
- N: N (placenta normally located) : pregnant women without suggestive signs of placenta previa or accreta on ultrasound
  Interventions: Diagnostic Test: serum BNP assessment

INTERVENTIONS:
Diagnostic Test: serum BNP assessment — serum BNP assessment in pregnant women with placenta previa, associated or not to a suspected abnormal placental invasion, compared to a control group

SUMMARY:
The placenta accreta is defined as a placenta that is abnormally adherent to the myometrium. It can thus invade the entire thickness of the myometrium (placenta increta) or even exceed the serosa and invade neighboring organs (placenta percreta). It is a rare obstetric pathology with significant morbidity, and its management most often requires hemostatic hysterectomy. Its frequency has increased significantly in recent decades due to the increased rate of caesareans.

The maternity center of Tunis ( CMNT ) is a level 3 maternity center, supporting over 12 000 births yearly, where the caesarean section's rate is very high, close to 45% of deliveries. Recently we noted an increase in abnormal placental invasion incidence : in 2018, we report over 60 cases of placenta accreta,increta and percreta.

Early detection of these patients can help reduce potential risks. Ultrasound and MRI are the main diagnostic tools, but each one has weaknesses. Biological approch of this diagnosis is not well studied. Recently, BNP has been shown to be associated with increased angiogenesis. Because placenta accreta is characterized by abnormal uteroplacental neovascularization, it has been hypothesized that serum BNP levels may be related to abnormal invasion of the placenta.

In the literature, only one study investigated the relationship between cardiac biomarkers (Pro-BNP, CK, CK-MB and troponins) and abnormalities of placental adhesion. The main conclusion was that the Pro-BNP could predict placental accretisation.

Thus, the BNP as a mean of screening, could enrich our diagnostic arsenal. The purpose of our study is to determine whether or not BNP can predict abnormal placental invasion during pregnany.

DETAILED DESCRIPTION:
The investigators will conduct a monocentric , prospective, observational study, including 60 pregnant women, with history of at least one previous uterine scar, and scheduled for cesarian delivery. The participants will be divided into 3 equal groups according to the imaging data obtained by a senior ultrasonographer , and the MRI data when necessary :

Ultrasonography will be performed in all participants. If placenta previa is diagnosed, without any suggestive signs of abnormal placental invasion, the patient is assigned to group P.

If placenta previa is diagnosed, and associated to suggestive signs of abnormal placental invasion,the patient is assigned to group I and an MRI will be performed.

If the ultrasonography is free of any suggestive signs of placenta previa, the patient is assigned to group N.

Finally :

* group P : pregnant women with placenta previa on ultrasound and no suggestive signs of abnormal placental invasion
* group I : pregnant women with placenta previa on ultrasound, and suggestive signs of abnormal placental invasion on ultrasound .
* group N : pregnant women without suggestive signs of placenta previa or abnormal placental invasion on ultrasound

After written and informed consent are obtained, a standard battery of blood tests including serum BNP will be runned.

For every patient, the following will be recorded : anthropometric measurements, previous obstetric and medical history, emergency or elective surgery, anesthetic technique, per-operative findings (placenta previa, placenta previa with abnormal placental invasion (accreta, increta, percreta), placenta normally located), amount of blood products transfused, nature of haemostasis procedures, complications.

Patients will be excluded, if their condition may cause a rise in serum BNP during the sample collection, those being: preterm premature rupture of membranes, acute anaemia or metrorrhagia, active labor, severe infections, arterial hypertension, known pulmonary hypertension, symptoms of heart failure, known hypertrophic or restrictive cardiomyopathy, history of valvular or congenital heart disease, atrial and ventricular tachyarrhythmias, pulmonary embolism, chronic obstructive pulmonary disease, kidney failure or renal dysfonction, liver dysfonction, severe metabolic and hormone abnormalities ( thyrotoxicosis or diabetic ketosis ), drug use possibly affecting cardiovascular system ( beta-blocker or other cardiovascular drug).

ANESTHETIC MANAGEMENT:

The timing of delivery is usually between 36 and 37 weeks for group P and I, and after 38 weeks for group N.

General anesthesia will be performed in pregnant women from group I and P. Regional anesthesia will be performed in pregnant women from group N.

Hemodynamic management during anesthesia for group I will require placement of 2 peripheral large-bore venous access, a desilet catheter in the femoral vein, and an arterial line preoperatively.

In patients from group P, 2 peripheral large-bore venous access will be placed preoperatively. A desilet catheter and arterial line will be obtained if necessary upon the anesthesiologist judgment.

In patients from group N, 1 peripheral large-bore venous access will be placed prior to the beginning of surgery.

Blood transfusion requirements will be based on the hemodynamic status, the amount of blood loss, the need of catecholamines and the anesthesiologist's experience.

Peroperatively, final diagnosis will be made according to surgical findings. If placenta is completely and easily removed, the diagnosis of abnormal placental invasion will not be retained.

If placenta could not be easily and completely removed, the diagnosis of abnormal placental invasion in established, and the case is carried out according to our surgical and anesthetic standards of management.

After collecting all groups, blood samples will be analysed for BNP, in a unique serie of tests.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with suspected placenta accreta on ultrasound or MRI
* pregnant women with suspected placenta previa on ultrasound or MRI
* pregnant women without sugestive signs of placenta previa or accreta on ultrasound
* history of at least one previous uterine scar
* written and informed consent

Exclusion Criteria:

* Preterm premature rupture of membranes
* Acute anaemia or metrorrhagia
* Active labor
* Severe infections
* Arterial hypertension
* known Pulmonary hypertension
* Symptoms of heart failure
* Known hypertrophic or restrictive cardiomyopathy
* History of valvular or congenital heart disease
* Atrial and ventricular tachyarrhythmias
* Pulmonary embolism
* Chronic obstructive pulmonary disease
* kidney failure or renal dysfonction
* Liver dysfonction
* Severe metabolic and hormone abnormalities ( thyrotoxicosis or diabetic ketosis )
* drug use possibly affecting cardiovascular system ( beta-blocker or other cardiovascular drug)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 60 parturients free from any exclusion criteria , devided equally into 3 groups :
  * group P : parturients with placenta previa on ultrasound and no suggestive signs of placenta accreta
  * group A : parturients with placenta previa on ultrasound, and suggestive signs of placenta accreta on ultrasound and / or MRI
  * group C : parturients without suggestive signs of placenta previa or accreta on ultrasound
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
serum BNP level | from the suspected diagnosis to study completion : up to 5 months
  compare BNP levels between group P ,I and N and compute serum BNP specificity and sensitivity in the detection of abnormal placental invasion

SECONDARY OUTCOMES:
blood loss | from the beginning of cesarean section to bleeding control : up to 48 hours
  compare the amount of blood loss in group P,I and N
blood transfusion | from the beginning of cesarean section to achieving hemodynamic stability : up to 48 hours
  compare blood transfusion requirements in group P,I and N

CONTACTS AND LOCATIONS:
Overall Officials: Hayen Maghrebi, PROFESSOR, Study Chair — University Tunis El Manar
Locations (1):
- Tunis maternity and neonatology center, minisetry of public health, Tunis, Tunisia